CLINICAL TRIAL: NCT01121809
Title: Plasma and Intracellular Concentrations of Raltegravir and Etravirine Administered Once Daily (800 mg and 400 mg, Respectively) Compared With Standard Dosing (400 mg and 200 mg/12 h) in Patients With HIV Infection
Brief Title: Plasma and Intracellular Concentrations of Raltegravir and Etravirine Administered Once Daily
Acronym: RAET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Luis Fernando Lopez-Cortes, Hospitales Universitarios Virgen del Rocío
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LLC-RAET-2009-1; 2009-014480-39 (EudraCT Number)
Record Dates: First submitted 2010-05-04; First posted 2010-05-12 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: Raltegravir; etravirine; pharmacokinetics; intracellular
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Other): Raltegravir 400 mg bid
  Interventions: Drug: Raltegravir
- Etravirine (Other): Etravirine 200 mg bid
  Interventions: Drug: Etravirine

INTERVENTIONS:
Drug: Raltegravir — Changing the dose of raltegravir from 400 mg bid to 800 mg qd
  Arms: Raltegravir
Drug: Etravirine — Changing the dose of etravirine from 200 mg bid to 400 mg qd
  Arms: Etravirine

SUMMARY:
Hypothesis: the intracellular concentrations of raltegravir (RAL) and etravirine (ETV) administrated as 800 and 400 mg once a day, respectively, are similar to those obtained with the standard doses of 400 and 200 mg/12h, respectively.

Objective: To analyze the plasma and intracellular concentrations of RAL and ETV administrated as 800 and 400 mg once daily respectively compared with standard doses of 400 and 200 mg/12h, respectively, and if they support its once daily administration.

DETAILED DESCRIPTION:
Objective: To analyze the plasma and intracellular concentrations of RAL and ETV administrated as 800 and 400 mg once daily respectively compared with standard doses of 400 and 200 mg/12h, respectively, and if they support its once daily administration.

Method: Phase IV, prospective, open labelled clinical trial with a planned duration of 24 weeks in which 16 patients from Hospitales Universitarios Virgen del Rocío will be enrolled. A 12 hours pharmacokinetic profile (immediately before and after 1, 2, 3, 4, 6, 8, 10 and 12 h) will be obtained after a supervised drug intake while taking RAL or ETV bid. Afterwards,the patients will take RAL or ETV once a day for 7 - 10 days. Subsequently, a new pharmacokinetic profile (predose and after 1, 2, 3, 4, 6, 8, 10, 12, 16, 20 and 24 h after a supervised drug intake) will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV-1-infected patients taking raltegravir- or etravirine-based antiretroviral regimens

Exclusion Criteria:

* Pregnancy
* Concomitant use of drugs that have potential interactions with raltegravir or etravirine pharmacokinetics
* Cirrhosis with clinical or analytic data of liver failure.
* Clinical history suggesting malabsorption or presence of diarrhea (> 3 stools / day) that could interfere with the absorption of study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in pharmacokinetic parameters (Cmax, Cmin, AUC, t1/2, and Cl), both in plasma and intracellular, of RAL and ETV. | baseline and 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, ND, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospitales Universitarios Virgen del Rocio, Seville, Sevilla, Spain

REFERENCES:
- [Derived] Gutierrez-Valencia A, Martin-Pena R, Torres-Cornejo A, Ruiz-Valderas R, Castillo-Ferrando JR, Lopez-Cortes LF. Intracellular and plasma pharmacokinetics of 400 mg of etravirine once daily versus 200 mg of etravirine twice daily in HIV-infected patients. J Antimicrob Chemother. 2012 Mar;67(3):681-4. doi: 10.1093/jac/dkr534. Epub 2011 Dec 21. PMID 22190606